CLINICAL TRIAL: NCT02314260
Title: Bishop Score; Are Further Modifications Needed?
Brief Title: Modifying Cervical Bishop Scoring System
Status: Completed | Type: Observational
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed M.Kamel, Lecturer Of obstetrics & Gynecology, Kasr El Aini Hospital
Other Study IDs: A13802022
Record Dates: First submitted 2014-12-06; First posted 2014-12-11 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Failed Induction of Labor
Keywords: labour induction; cervical length; trans-vaginal assessment of cervical length; Bishop score
MeSH Terms: interventions — Labor, Induced

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Labour Induction: 80 primigravidas undergoing bishop score calculation, trans-vaginal ultrasound assessment of cervical length &, Modified bishop score calculation, then induction of labour at our hospital.
  Interventions: Other: bishop score calculation; Other: Trans-vaginal ultrasound; Other: Modified bishop score calculation; Procedure: labour induction

INTERVENTIONS:
Other: bishop score calculation — Assessment of bishop score by vaginal examination
Other: Trans-vaginal ultrasound — trans-vaginal ultrasound assessment of cervical length.
Other: Modified bishop score calculation — using the cervical length and the original bishop score to calculate modified bishop score
Procedure: labour induction — Induction of labor was carried out as per our hospital's standard protocol.

SUMMARY:
To have an early more precise way to predict failed induction in patients undergoing elective termination of pregnancy & those more likely to undergo caesarian section,this will Spare patients with decreased chances of favorable induction a long and exhausting trial of labour with increased probability of complications and an emergency caesarian

DETAILED DESCRIPTION:
After approval of the ethical & scientific committees of the OBGYN department of Kasr El Aini hospital, 80 primigravidas undergoing induction of labour at our hospital in a prospective blind study were subjected to history taking, examination, investigations & ultrasonography. Indication for pregnancy termination was explained to each patient and a written consent was obtained.

Clinical examination & assessment:

Patients were examined vaginally by the attending physician and a Bishop score was assigned and recorded according to the original bishop scoring system 1964 (Bishop EH, 1964) as seen in table 1.

Table 1: The Bishop score (Bishop EH, 1964):

0 points : for no dilation, effacement 0-30%, station -3, firm consistency & posterior position of cervix

1. point : for dilation 1-2 cm, effacement 40-50%, station -2, medium consistency & mid position of cervix.
2. points: for dilation 3-4 cm, effacement 60-70%, station -1, soft consistency & Anterior position of cervix.
3. points: for dilation 5-6 cm, effacement 80%, station +1 or +2.

Sum of the points in each criteria assessed will be the bishop score.

Trans-vaginal ultrasound assessment of cervical length was performed using the same machine each time Sonoace x4 (samsung Medison Co., Ltd. Seoul, South Korea) following a standardized technique in which the bladder was emptied & the vaginal probe 6.5MHz was introduced into the vagina and manipulated so that the main anatomical landmarks (bladder, fetal presentation, cervical canal, internal and external cervical os) were identified. The hyper echoic line extending from the internal os to external os, was identified by fine manipulations of the probe. The cervical canal length was measured as the distance between the internal and external os, while presence of funneling was recorded. Funneling was defined as a (V)or (U) shaped indentation of the internal os. In the presence of funneling, the length of an associated funnel was not included as part of the cervical length, and the measurement was taken from the apex of the funnel to the external os.

A modified bishop score was devised for the purpose of this study, which aimed to incorporate cervical length into the bishop scoring system. This score was calculated by addition or subtraction of the figure obtained respectively for cervical length in table 2 from the original bishop score.

Table 2: Scoring System for respective cervical length

Score: -2 for Cervical length > 2.5cm by trans-vaginal ultrasound. Score: -1 for Cervical length 2 - 2.5 cm by trans-vaginal ultrasound.

Score: 0 for Cervical length 1.6 - 1.9 cm by trans-vaginal ultrasound.

Score: +1 for Cervical length 1 - 1.5 cm by trans-vaginal ultrasound.

Score: +2 for Cervical length < 1 cm by trans-vaginal ultrasound.

We think an unfavorable score should decrease the value of the bishop score, and not just fail to increase it (in comparison to the original score) & hence our negative value for unfavorable cervical length. The values used to set the figures for the max and min score for cervical length in table 2 were based on our observation of how several studies displayed the range of their results for cervical length and how we think that it should impact the bishop score. There is no exact pre-set cut off value for what a favorable cervical length should be.

Labour induction and Monitoring:

Induction of labor was carried out as per our hospital's standard protocol, in which patients with unfavorable cervical examination i.e. bishop score of 4 or less were given dinoprostone 3mg (Dinoglandin E2 ® Egypharma Nasr City Cairo Egypt) vaginal tablet, with re-dosing intervals every six hours if no significant cervical changes were noted.

In cases where the initial bishop score was 5 or more, or improvement was seen after dinoprostone, Oxytocin was initiated for induction. In cases already having one or more dinoprostone vaginal tablets, oxytocin was started four hours after the final dinoprostone dose, using the low-dose protocol beginning with 2 mU/min (and increase by 2 mU/min) at incremental time intervals (15 - 30 minutes). The goal was to reach satisfactory contractions (3-5 per ten minutes with each contraction lasting 45 seconds), & to avoid uterine hyperstimulation.

All through induction & labor fetal heart rate was measured every 30 minutes in first stage of labor and every 10 minutes in second stage of labor. Progress of labor was observed & recorded, the total amount of oxytocin used, fetal weight and Apgar score for each baby were recorded. The total time taken till reaching active phase of labor, total time taken till delivery & mode of delivery were recorded. Any decision to proceed to caesarean was reviewed by a senior consultant and the indication was noted. Any case undergoing caesarean for any indication other than failure of progress will be omitted from the results.

ELIGIBILITY:
Inclusion Criteria:

1. Primigravida Singleton pregnancy with mature fetus at term indicated for termination of pregnancy.
2. Cephalic presentation.
3. Medical indications for termination of pregnancy e.g.: Pre-eclampsia, uncontrolled diabetes at term..e.t.c,
4. Post-term pregnancy.
5. Fetal indication: signs of fetal compromise e.g.: decreased biophysical profile, poor umbilical Doppler indices, diminished liquor.
6. premature rupture of membranes (PROM) not going into spontaneous labor within 24 hours since onset.
7. Intrauterine fetal death (IUFD).

Exclusion Criteria:

1. they had true labor pains or clear onset of labor as diagnosed by cervical changes.
2. Previous uterine surgery (scared uterus).
3. Cephalo-pelvic disproportion.
4. Mal-presentations
5. Severe oligo-hydramnios i.e.: amniotic fluid index Less than 5.
6. Twin pregnancy.
7. Fetal macrosomia. -Growth beyond a specific threshold (weight above 4000g) 8) Placenta previa.

9) Fetal bradycardia in case of living fetus.

Ages: 20 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 80 primigravidas undergoing induction of labour at our hospital in a prospective study were subjected to history taking, examination, investigations & ultrasonography. Indication for pregnancy termination was explained to each patient and a written consent was obtained.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Kamel, M.D, Principal Investigator — Lecturer of obstetrics & Gynecology
Locations (1):
- 11562, Ḩadā’iq al Qubbah, Cairo Governorate, Egypt

REFERENCES:
- [Background] BISHOP EH. PELVIC SCORING FOR ELECTIVE INDUCTION. Obstet Gynecol. 1964 Aug;24:266-8. No abstract available. PMID 14199536

RESULTS

PARTICIPANT FLOW:
Recruitment Details: started July 2014 till December 2014 & recruited 80 primigravidas undergoing scheduled for pregnancy termination at Kasr El Aini Hospital
Period: Overall Study
Arm/Group | Labour Induction
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 80 primigravidas undergoing induction of labour at our hospital
Arm/Group | Labour Induction
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.31 (3.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 0
Region of Enrollment [Number; unit: participants]
  Egypt | 80
Gestational Age [Mean (Standard Deviation); unit: Weeks] | 39.70 (1.50)
Bishop Score [Mean (Standard Deviation); unit: units on a scale] — A score of 5 or less suggests that labour is unlikely to start without induction. A score of 9 or more indicates that labour will most likely commence spontaneously.
  The score can range between (0 -13) A low Bishop's score often indicates that induction is unlikely to be successful, however there is no set value
  units on a scale | 5.71 (1.20)
Cervical Length [Mean (Standard Deviation); unit: Cm] | 2.06 (0.56)
New Modified Bishop Score [Mean (Standard Deviation); unit: units on a scale] — The modified bishop score, is tailored by criteria we added to incorporate cervical length into the old bishop score.
  it can have a range between (-2 & 15). low scores bellow 5 are associated with failed induction , while high scores are associated with successful vaginal delivery.
  there are no set cut-off value for failed induction
  units on a scale | 5.28 (1.88)
Time to active Phase [Mean (Standard Deviation); unit: Hours] | 11.87 (3.25)
Induction to delivery time [Mean (Standard Deviation); unit: Hours] | 17.38 (4.29)
rupture of membraned duration [Mean (Standard Deviation); unit: hours] | 9.93 (4.50)
Fetal weight (kilograms) [Mean (Standard Deviation); unit: kilograms] | 3.02 (0.267)
Apgar score at 5 minutes [Mean (Standard Deviation); unit: units on a scale] — Apgar score is a method to assess the health of a newborn immediately after birth.
  It is determined by evaluating the newborn baby on 5 simple criteria on a scale from 0-2, then adding the five values obtained.
  The resulting Apgar score ranges from 0-10. The 5 criteria are summarized using words chosen to form a backronym (Appearance,Pulse,Grimace,Activity,Respiration).
  The test is generally done at 1 & 5 minutes after birth. Scores 7 & above are normal, 4-6 fairly low,and 3 and below are critically low.A low score on the one-minute test, may indicate neonate requires medical attention
  units on a scale | 8.45 (1.82)

OUTCOME MEASURES:

1. Primary Outcome: Area Under Receiver Operating Characteristic Curve (ROC) for Modified Bishop Score
Description: to predict failed induction and comparing it to the area under curve for bishop score to find out which test is more accurate in predicting caesarean section, The positive actual state is failed induction and performing Caesarean Section.The positive actual state is failed induction, the true positive rate (Sensitivity) is plotted in function of the false positive rate (100-Specificity). So as the numbers approaches 1, induction fails, the Y-axis of the curve is sensitivity and the x- axis is (1-specificity).
Time Frame: 5 months
Population: the area under the modified bishop score was 0.916 (95% [confidence interval ] 0.85-0.97). The positive actual state is failed induction and performing Caesarean Section, So as the numbers approaches 1, induction fails, the Y-axis of the curve is sensitivity and the x- axis is (1-specificity).
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Labour Induction
Number analyzed (Participants) | 80
probability | 0.916 [0.85 to 0.97]
Statistical Analysis 1: Comparison: Labour Induction; Null hypothesis: true area = 0.5 The positive actual state is failed induction, the true positive rate (Sensitivity) is plotted in function of the false positive rate (100-Specificity); Test type: Superiority or Other; p = 0.000, t-test, 2 sided — Under the nonparametric assumption. P-value <0.05, means statistical significance; Mean Difference (Final Values) = 0.917, 95% CI 2-sided [0.854 to 0.979], Standard Error of Mean 0.0318 — The positive actual state is failed induction and performing Caesarean Section, So as the numbers approaches 1, induction fails. the Y-axis of the curve is sensitivity and the x- axis is (1-Specificity)

2. Secondary Outcome: Area Under Curve for The Bishop Score
Description: to predict failed induction and comparing it to the area under curve for modified bishop score to find out which test is more accurate in predicting caesarean section, The positive actual state is failed induction and performing Caesarean Section. The positive actual state is failed induction, the true positive rate (Sensitivity) is plotted in function of the false positive rate (100-Specificity), So as the numbers approaches 1, induction fails, the Y-axis of the curve is sensitivity and the x- axis is (1-specificity).
Time Frame: 5 months
Population: The positive actual state is failed induction and performing Caesarean Section, So as the numbers approaches 1, induction of labour fails, the Y-axis of the curve is (sensitivity) and the x- axis is (1-specificity).
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Labour Induction
Number analyzed (Participants) | 80
probability | 0.806 [0.69 to 0.91]
Statistical Analysis 1: Comparison: Labour Induction; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.000, t-test, 2 sided — Under the nonparametric assumption P value <0.05 is statistically significant; Mean Difference (Final Values) = 0.806, 95% CI 2-sided [0.693 to 0.919], Standard Error of Mean 0.0578 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Cut Off Value for The Modified Bishop Score
Description: the value at which there a high sensitivity and specificity to predict failed labour induction
Time Frame: 5 months
Population: sensitivity of 83% and a specificity of 87% for failed induction.
Measure: Number; unit: probability
Arm/Group | Labour Induction
Number analyzed (Participants) | 80
probability | 4.5
Statistical Analysis 1: Comparison: Labour Induction; The smallest cutoff value is the minimum observed test value minus 1, and the largest cutoff value is the maximum observed test value plus 1. All the other cutoff values are the averages of two consecutive ordered observed test values; Test type: Superiority or Other; p = 0.000, t-test, 2 sided — P<0.05 is significant; Slope = 4.5, 95% CI 2-sided [0.00 to 10], Standard Error of Mean 0.0318 — at a cutoff value of 4.5, the sensitivity for failure to labour induction is 0.83 (83%), with a specificity of 0.87(87%)

4. Secondary Outcome: Cut Off Value for Bishop Score
Description: the value at which there a high sensitivity and specificity to predict failed labour induction
Time Frame: 5 months
Population: sensitivity of 83% & specificity was 73% to failed induction
Measure: Number; unit: probability
Arm/Group | Labour Induction
Number analyzed (Participants) | 80
probability | 5.5
Statistical Analysis 1: Comparison: Labour Induction; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.000, t-test, 2 sided — P<0.05 is significant; Mean Difference (Final Values) = 5.5, 95% CI 2-sided [0.00 to 10], Standard Error of Mean 0.0578 — at a cutoff value of 5.5, the sensitivity for failure to labour induction is 0.83 (83%), with a specificity of 0.73 (73%)

ADVERSE EVENTS:
Time Frame: 5 months. total time to complete study, other adverse events not related to successful labour induction were not recorded e.g postpartum hemorrhage, wound infection e.t.c
Description: In our study the only serious adverse event recorded was Caesarean section, which occurred when labour progress stopped,& labour induction was considered to be a failure. In the 5 months total time to complete study, other adverse events not related to successful labour induction were not recorded e.g postpartum hemorrhage, wound infection e.t.c
Arm/Group | Labour Induction
Serious Adverse Events (participants affected / at risk) | 18/80
Other Adverse Events (participants affected / at risk) | 0/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Labour Induction (N=80)
failed labour induction (Pregnancy, puerperium and perinatal conditions) | 18 — caesarean section was performed due to failed progress of labour

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes